CLINICAL TRIAL: NCT03431636
Title: Effect of Different Techniques of Recovery After Fadiga in Para-athletes
Brief Title: Effect of Different Techniques of Recovery in Para-athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, first investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fadiga in para-athletes
Record Dates: First submitted 2017-12-18; First posted 2018-02-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pain; Recruitment
Keywords: sports for people with disabilities; immersion therapy; cryotherapy; physiotherapy
MeSH Terms: conditions — Pain | interventions — Immersion; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersion in cold water (Experimental): The athlete will remain submerged in a "Cryo Control - Ice Bath Systems®" bathtub, which allows filtration and maintenance of constant water temperature, and shoulder blade water (Getto and Golden, 2013) for 15 minutes in the 15 degrees Celsius (Machado et al, 2016).
  Interventions: Other: immersion
- Ice pack (Active Comparator): The athlete will remain for 20 minutes with plastic packets of 500 grams of ice each, in the region of the evaluated muscles.
  Interventions: Other: ice pack
- Control (Sham Comparator): Group in which the athlete will be instructed to remain seated in a comfortable position, at rest, for 20 minutes.
  Interventions: Other: rest

INTERVENTIONS:
Other: immersion — cold water immersion
  Arms: Immersion in cold water
Other: ice pack — ice packs through the body
  Arms: Ice pack
Other: rest — seated rest
  Arms: Control

SUMMARY:
Para-athletes are submitted and intense efforts in training and competitions that often overlap in days and weeks. In this sense, and in the search for better brands and indexes, it is necessary to use recovery methods that allow less late muscle pain and better physical performance. Recovery methods are widely used in athletes of various modalities, however there are no studies that point out their effects on para-athletes. This highlights the need for studies on this topic. Paragliding athletes, who train at the Londrina Yacht Club, Londrina Canoeing and Rowing School, who present paraplegia after spinal cord injury, with motor level T10 or lower, without any problem of thermoregulation will participate in the study. All were male and female, with no complaints of musculoskeletal pain or history of upper limb muscle injuries in the last six months and with the same demand for training and competitions. Initially an evaluation will be performed where 1RM, VO2 max, pain, spasticity, body temperature, heart rate variability and electromyographic signal of the involved muscles will be tested. After three days they will be induced to fatigue through a protocol in the traction exercise and immediately directed to one of the 3 intervention groups: ice pack, immersion in cold water or rest. The same baseline evaluations will be repeated after 24, 48 and 72 hours. It is expected that the group submitted to immersion in cold water presents better parameters for pain and sports performance.

DETAILED DESCRIPTION:
Athletes who agree to participate in the study will sign the ICF and will respond to the questionnaire to characterize the sample. All procedures will be carried out at the Londrina Canoeing and Rowing School, where athletes are trained.

In the sequence the athlete will be submitted to the test of a maximum repetition (1RM) of the exercise of traction with the upper limbs, which is specific for canoeing.

This will be performed with the athlete positioned in a decubitus position and well positioned. In the following, it will be advised to lift the bar with load determined by the athlete as adequate to carry out the movement, in case of carrying out the movement with ease and without compensations of other parts of the body the load will increase until the athlete is no longer able to perform the movement with quality, and then the maximum load determined as the one in which it was able to perform the complete movement for the last time.

On the first day of collection, the maximum VO2 test will be performed, where the athlete will perform a test of 8 to 12 minutes where a progressive load will be introduced until the athlete reaches his maximum oxygen consumption and is no longer able to continue the test.

After three days the athlete will return to the collection site to perform the tests in three moments:

1. At rest (lying supine on a stretcher):

   * HR variability
   * VO2
   * Resting body temperature
   * Assessment of spasticity by the Ashworth scale
   * Borg Fatigue Scale.
   * EVA
   * pressure pain threshold (LDP)
2. During simulation of the paddle on the K1 ergometer (figure 2), which will be held for 6 minutes at comfortable pace, where the last minute data will be used:

   * IN G
   * VO2
   * HR variability After the end of the evaluations, the athlete will be submitted to the fatigue protocol where he will be guided, to perform the maximum movements of the traction exercise with load referring to 60% of the 1RM, twice, with interval of 1 minute between them.

Then it will be taken to another place, near the collection room for randomization, by means of a draw in a sealed and opaque envelope in one of the three study groups:

* Cold water immersion: The athlete will remain submerged in a "Cryo Control - Ice Bath Systems®" bathtub, which allows filtration and maintenance of constant water temperature, and shoulder blade water for 15 minutes in the water at 15 degrees Celsius.
* Ice pack: The athlete will remain for 20 minutes with plastic packets of 500 grams of ice each, in the region of the evaluated muscles.
* Control: Group in which the athlete will be instructed to remain seated in a comfortable position, at rest, for 20 minutes.

The randomization and execution of the protocols will be carried out in environments that the evaluators do not have vision or access, to favor the blindness of the evaluations.

After termination of the intervention protocol, the athlete will be instructed to maintain routine sleep and feeding activities with the rest of the team, but without participation in any type of training or physical activity for the next 3 days.

ELIGIBILITY:
Inclusion Criteria:

* paraplegia after spinal cord injury, with motor level T10 or lower, without any problem of thermoregulation
* athletes of the modality paracanoagem, that train in the Yacht Club of Londrina, in the School of canoagem and rowing of Londrina

Exclusion Criteria:

* cold allergies
* upper limb surgery in the last six months
* scarring or skin lesions
* peripheral vascular perfusion abnormalities
* viral conditions (such as colds or flu)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-07-25 (Estimated); Primary Completion 2020-10-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
evolution of muscular pain | pre, immediately after, after 24, 48 and 72 hours
  late muscle pain will be assessed at various times to detect changes caused by fatigue will be analyzed through the threshold of pressure pain, in view of the induction of pain caused to the study, the pain will be monitored at various times

SECONDARY OUTCOMES:
oxygen consumption | pre, immediately after, after 24, 48 and 72 hours
  will be analyzed the percentage of maximum VO2 used for a given task by means of gas analyzer
spasticity | pre, immediately after, after 24, 48 and 72 hours
  by ashworth scale
muscle recruitment | pre, immediately after, after 24, 48 and 72 hours
  with electromyography during rowing task
heart rate variability | pre, immediately after, after 24, 48 and 72 hours
  by polar, during the paddling activity

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, Principal Investigator — State University of Londrina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price MJ. Thermoregulation during exercise in individuals with spinal cord injuries. Sports Med. 2006;36(10):863-79. doi: 10.2165/00007256-200636100-00005. PMID 17004849
- [Background] Ihsan M, Watson G, Abbiss CR. What are the Physiological Mechanisms for Post-Exercise Cold Water Immersion in the Recovery from Prolonged Endurance and Intermittent Exercise? Sports Med. 2016 Aug;46(8):1095-109. doi: 10.1007/s40279-016-0483-3. PMID 26888646